CLINICAL TRIAL: NCT04525274
Title: Comparative Study Between Intraperitoneal Dexmedetomidine Versus Ketamine With Bupivacaine For Postoperative Analgesia After Laparoscopic Sleeve Gastrectomy
Brief Title: Intraperitoneal Dexmedetomidine Versus Ketamine With Bupivacaine For Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rehab Abd-Allah Wahdan, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-7-2020
Record Dates: First submitted 2020-08-16; First posted 2020-08-25 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Obesity
Keywords: sleeve gastrectomy; postoperative analgesia; intraperitoneal dexmedetomidine; intraperitoneal ketamine
MeSH Terms: conditions — Obesity | interventions — Saline Solution; Dexmedetomidine; Ketamine

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three equal groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: triple blinded (patient, surgeon and outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): patient will receive 40 ml bupivacaine 0.25% + 5 ml normal saline with a total volume of 45 ml to be installed intraperitoneally.
  Interventions: Drug: normal saline
- dexmedetomidine group (Active Comparator): patient will receive 40 ml bupivacaine 0.25% + 1 µg/kg dexmedetomidine diluted in 5 ml normal saline with a total volume of 45 ml to be installed intraperitoneally.
  Interventions: Drug: dexmedetomidine
- ketamine group (Active Comparator): patient will receive 40 ml bupivacaine 0.25% + 0.5 mg/kg ketamine diluted in 5 ml normal saline with a total volume of 45 ml to be installed intraperitoneally.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: normal saline — At the end of surgery, patient will be shifted to Trendelenburg position and intraperitoneal instillation of 40 ml bupivacaine 0.25% + 5 ml normal saline will be done guided by the camera and sprayed uniformly into the peritoneal cavity by the surgeon.
  The patient will be maintained in Trendelenburg position for 5-10 minutes after drug instillation and the abdomen will be deflated by passive exsufflation using gentle abdominal pressure.
  Arms: control group
Drug: dexmedetomidine — At the end of surgery, patient will be shifted to Trendelenburg position and intraperitoneal instillation of the study drug(40 ml bupivacaine 0.25% + 1 µg/kg dexmedetomidine diluted in 5 ml normal saline) will be done guided by the camera and sprayed uniformly into the peritoneal cavity by the surgeon.
  The patient will be maintained in Trendelenburg position for 5-10 minutes after drug instillation and the abdomen will be deflated by passive exsufflation using gentle abdominal pressure.
  Arms: dexmedetomidine group
Drug: Ketamine — At the end of surgery, patient will be shifted to Trendelenburg position and intraperitoneal instillation of the study drug(40 ml bupivacaine 0.25% + 0.5 mg/kg ketamine diluted in 5 ml normal saline) will be done guided by the camera and sprayed uniformly into the peritoneal cavity by the surgeon.
  The patient will be maintained in Trendelenburg position for 5-10 minutes after drug instillation and the abdomen will be deflated by passive exsufflation using gentle abdominal pressure.
  Arms: ketamine group

SUMMARY:
Post-laparoscopic sleeve pain management is essential for early mobilization of the patient and so on decrease post-operative complication. The use of opioids is associated with adverse effects such as nausea, pruritus, sedation, and occasionally respiratory depression.

Previous studies stated that intraperitoneal instillation of bupivacaine alone has been used to reduce acute postoperative abdominal and shoulder pain allow early mobilization and decrease postoperative opioid requirements and its complications.

In this study the investigators will compare between intraperitoneal instillation of dexmedetomidine with bupivacaine versus ketamine with bupivacaine in patients undergoing laparoscopic sleeve gastrectomy under general anesthesia regarding to postoperative pain relief to reduce morbidity and mortality.

DETAILED DESCRIPTION:
Obesity is a serious condition in developed and developing countries occur due to some hormonal disorder or due to reduce energy expenditure with increasing energy uptake [1]. Nowadays, obesity considered the second cause of deaths after smoking all over the world [2].

Severe obesity increase the incidence of many chronic disease such as (diabetes mellitus, hypertension, cardiovascular diseases and others) [3]. This leads to substantial morbidity, early mortality [4], impaired quality of life [5] and excess healthcare expenditures [6].

Laparoscopic bariatric surgery is the most recommended and effective long-term treatment for morbid obesity (which body mass index (BMI) ≥40 kg/m2) and obesity-related complication [7].

Postoperative pain management after laparoscopic sleeve still considers a major challenge. As many of the patients express moderate-to-severe pain in postoperative period [8]. Causes of postoperative pain include inflammation of the peritoneum, intra-abdominal cavity stretch and irritation of diaphragm by carbon-dioxide (CO2) remains in the abdominal cavity [9].

Multimodal analgesia regimens such as parenteral opioids, nonsteroidal anti-inflammatory drugs and intraperitoneal instillation of different drugs such as local anesthetic drugs alone or with adjuvants like; opioid and α2 agonists' drugs such as clonidine and dexmedetomidine have been tried to reduce overall pain and postoperative complications of patients undergoing laparoscopic surgeries [8, 9].

Bupivacaine is the most commonly used local anesthetic drug, its intraperitoneal instillation has become a popular practice for pain relief after laparoscopic surgery as it causes blockade of free afferent nerve endings in peritoneum [10].

Dexmedetomidine, the pharmacologically active d-isomer of medetomidine, it is a potent and highly selective α2-adrenoreceptor agonist with sympatholytic, sedative, amnestic, anxiolytic, neuroprotective and analgesic properties [11].

Ketamine is an immunomodulatory agent and anti-inflammatory drug and it has a noncompetitive antagonist of the N-methyl-d-aspartate (NMDA) receptor that blocks nociceptive input and reduce hyperalgesia [12].

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age 21-60 years old.
* Sex both male and female.
* BMI ≥40 kg/m2
* ASA II and ASA III.
* Scheduled for elective laparoscopic sleeve gastrectomy under general anesthesia.

Exclusion Criteria:

* Patients with known history of allergy to study drugs.
* Patients with uncontrolled diabetes mellitus.
* Psychological and mental disorders.
* Severe hypertensive, cardiac, hepatic and renal patients.
* Patients on opioid or sedative use.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
change in assessment of postoperative shoulder, abdominal and incisional pain | at 1, 2, 4, 6, 12 and 24 hours postoperatively
  will be assessed by visual analogue scale (VAS) scale, On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain.

SECONDARY OUTCOMES:
Time of first request of analgesia | within 24 hour postoperative
  time elapsed from patient arrival to PACU [T0] to time of first patient call for analgesia
Total rescue analgesic requirement | during the first postoperative 24 hours
  if VAS ≥3 or on patient request, rescue analgesia will be given
The incidence of postoperative nausea and vomiting (PONV) | during the first postoperative 24 hours
  occurrence of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Result] Ozkan AS. Anesthesia management in sleeve gastrectomy: Single center experience. Annals of Medical Research. 2018; 25(4)613-8.
- [Result] Tekeli AE, Eker E, Bartin MK, Oner MO. Anesthesia Management in Laparoscopic Sleeve Gastrectomy Cases. East J Med. 2019; 24(3): 335-9.
- [Result] Praveena BL, Bharathi B, Sahana VR. Intraperitoneal Ropivacaine with Dexmedetomidine or Fentanyl for Postoperative Analgesia Following Laparoscopic Cholecystectomy: A Comparative Randomized Trial. Anesth Essays Res. 2019 Jan-Mar;13(1):169-173. doi: 10.4103/aer.AER_191_18. PMID 31031500
- [Result] Beder El Baz MM, Farahat TEM. Intraperitoneal Levobupivacaine Alone or with Dexmedetomidine for Postoperative Analgesia after Laparoscopic Cholecystectomy. Anesth Essays Res. 2018 Apr-Jun;12(2):355-358. doi: 10.4103/aer.AER_205_17. PMID 29962597
- [Result] EL-Gaby SS, Mohammed SS. Intraperitoneal ketamine attenuates the inflammatory reactivity associated with pneumoperitoneum. Research and Opinion in Anesthesia & Intensive Care. 2017; 4:149-55.